CLINICAL TRIAL: NCT01814332
Title: CRF Receptor Antagonist for PTSD and Related Sleep Disturbances in Women
Brief Title: Analyzing Female Trauma Exposed Responses to a Medication
Acronym: AFTER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09S-NIMH-002
Record Dates: First submitted 2013-03-11; First posted 2013-03-19 (Estimated); Results first posted 2016-04-25 (Estimated); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Stress Disorders, Post-traumatic
Keywords: Stress disorders, Post-traumatic; Sleep
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — NBI 77860; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- GSK561679 (Experimental): GSK561679, oral administration, 350mg/day, 6 week administration
  Interventions: Drug: GSK561679
- Placebo (Placebo Comparator): Placebo compound treatment for comparison with IP
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK561679 — GSK561679, oral administration, 350mg/day, 6 week administration
  Other Names: CRF1 antagonist
  Arms: GSK561679
Drug: Placebo — Placebo compound treatment for comparison with IP
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
This purpose of this study is to look at the safety of the experimental drug GSK561679 as well as its effects on PTSD symptoms, thinking and memory, startle reaction, stress hormones, and mental health symptoms in comparison to placebo (an inactive substance).

DETAILED DESCRIPTION:
A growing body of literature suggests that stress-related disorders such as PTSD are associated with chronically increased activity of CNS circuits that utilize corticotropin-releasing factor (CRF), a neuropeptide involved in mediating the neuroendocrine, immune, autonomic, and behavioral responses to stress. CRF1 receptor antagonists exert significant dampening effects on this system, but have never been investigated in patients with PTSD. The investigators at Mount Sinai School of Medicine (MSSM) and the National Institute of Mental Health (NIMH) Intramural Research Program have conducted a Phase II proof-of-concept clinical trial of a neurokinin-1 antagonist provided by GlaxoSmithKline (GSK). In this investigation, we will conduct a 2-site (Emory and MSSM), 6-week, randomized, double-blind, placebo-controlled, parallel-arm, fixed dose trial evaluating the efficacy, safety, and tolerability of GSK561679 for 154 female adult outpatients with PTSD. The San Francisco Department of Veterans Affairs Medical Center (SFVAMC) was added as a site in July 2012. SFVAMC will enroll 40 female adult outpatients with PTSD.

We propose to investigate the efficacy of the highly specific CRF1 antagonist GSK561679 in PTSD in a placebo-controlled clinical trial. GSK561679 has not been approved by the Food and Drug Administration for the treatment of any condition. Furthermore, we propose to longitudinally investigate whether certain biological surrogate markers (neuroendocrine, neurophysiology, genotyping) are predictive of treatment response. If a patient is already taking medication for PTSD and has achieved therapeutic response, she will not be tapered off effective medication(s) to participate in this study, and will not be eligible for the study. Taper and discontinuation of medications in preparation for this study will only occur in those patients who are not responding to medication treatment for PTSD.

Preclinical and clinical literature also exists which implicates both hypothalamic and extra hypothalamic CRF in stress-related insomnia and the regulation of non-rapid eye movement delta sleep. There is preliminary evidence that blocking CRF signaling results in an immediate improvement in stress-related sleep disturbances. Disturbed sleep is the most prevalent symptom endorsed by PTSD patients. It is potentially debilitating in many domains of functioning, and it is an outcome that can be objectively and precisely measured with sleep EEG. Therefore, an exploratory aim of this study will be to investigate the impact of GSK561679 on objective measures of sleep continuity and quantitative sleep EEG using ambulatory polysomnography. All subjects enrolled at SFVAMC who meet inclusion and exclusion criteria for the study will be given the option of having their sleep monitored throughout the study

ELIGIBILITY:
Inclusion Criteria:

* Female between 18-65 years of age
* Able to provide consent and willing to participate in research
* PTSD duration of illness at least 3 months
* Negative Urine toxicology test
* Agrees to use protocol-defined effective birth control method

Exclusion Criteria:

* Subject is currently participating in another clinical trial in which she is or will be exposed to an investigational or non-investigational drug or device, or has done so within the preceding month for studies unrelated to PTSD, or 1 month for studies related to PTSD
* Subject has a documented history of hepato-biliary disease including a history of, or positive laboratory results for hepatitis
* Subject requires ongoing treatment with medications that are prohibited per protocol
* Subject has a stool positive for occult blood.
* Pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 128 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2014-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C. Neylan, MD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (1):
- San Francisco VA Medical Center, San Francisco, CA, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Emory University School of Medicine, Mount Sinai School of Medicine, Baylor College of Medicine, and the San Francisco VA Medical Center between January 2010 and June 2014.
Pre-assignment Details: Subjects stopped psychotropic medications (w/ the exception of zolpidem, eszopiclone, and zaleplon for insomnia) w/in 2 weeks (6 weeks for fluoxetine) of Visit 1. Patients on ineffective psychotropic medications tapered off by the patients' prescribing doctor. 150 subjects did not proceed to randomization due to meeting exclusionary criteria.
Period: Overall Study
Arm/Group | GSK561679 | Placebo
Started | 63 | 65
Completed | 47 | 49
Not Completed | 16 | 16
Not completed — Adverse Event | 8 | 3
Not completed — Withdrawal by Subject | 3 | 8
Not completed — Protocol Violation | 0 | 4
Not completed — Lost to Follow-up | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK561679 | Placebo | Total
Number analyzed (Participants) | 63 | 65 | 128
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 63 | 65 | 128
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 65 | 128
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 63 | 65 | 128

OUTCOME MEASURES:

1. Primary Outcome: Efficacy, Measured by Change in the Clinician-Administered PTSD Scale (CAPS) Score
Description: The CAPS is a semi-structured clinical interview providing a measure of the severity of PTSD symptoms. A severity score is calculated by summing the frequency and intensity scores for each of the 17 DSM-IV criteria symptoms. The severity of symptoms is rated on a scale from 0-4, where, 0 = Absent, 1 = Mild/subthreshold; 2 = Moderate/ threshold, 3 = Severe/markedly elevated and 4 = Extreme/ incapacitating. Scores may range from 0 (no symptoms) to 136 (severe symptoms). Change is the difference in scores between baseline and 6 weeks.
Time Frame: Baseline, 6 weeks
Population: Intent to treat analysis was performed using maximum likelihood estimation with mixed models to include all observations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 63 | 65
score on a scale | -26.02 (22.28) | -27.33 (19.76)

2. Secondary Outcome: Efficacy, Measured by Response Rate of at Least 50% Improvement in CAPS Score at the End of 6 Weeks as Compared to Baseline
Description: The number of participants that showed at least a 50% reduction in CAPS scores from their baseline visit at the end of 6 weeks were measured as having a response to the treatment. The CAPS is a semi-structured clinical interview providing a measure of the severity of PTSD symptoms. A severity score is calculated by summing the frequency and intensity scores for each of the 17 DSM-IV criteria symptoms. Scores may range from 0 (no symptoms) to 136 (severe symptoms).
Time Frame: Baseline, Week 6
Measure: Number; unit: participants
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 63 | 65
participants | 14 | 18

3. Secondary Outcome: Efficacy, Measured by Change in the Montgomery-Asberg Depression Rating Scale (MADRS) Score
Description: The MADRS is a ten-item clinician-administered questionnaire used to measure the severity of depressive symptoms in patients with depressive disorders. Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60. Change is the difference in scores between baseline and 6 weeks.
Time Frame: Baseline, Week 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 63 | 65
Score on a scale | -7.83 (9.32) | -5.98 (9.10)

4. Secondary Outcome: Safety, Measured by the Number of Subjects That Experienced an Adverse Event
Description: The occurrence of adverse events will be recorded at the end of 6 weeks.
Time Frame: Baseline, Week 6
Measure: Number; unit: participants
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 63 | 65
participants | 55 | 55

ADVERSE EVENTS:
Arm/Group | GSK561679 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/63 | 1/65
Other Adverse Events (participants affected / at risk) | 55/63 | 55/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK561679 (N=63) | Placebo (N=65)
Anaphylaxis (Immune system disorders) | 0 (0) | 1 (1) — Anaphylactic reaction to seafood in person with known allergy to seafood
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK561679 (N=63) | Placebo (N=65)
Tinnitus (Ear and labyrinth disorders) | 3 (3) | 0 (0)
Hot Flush (Endocrine disorders) | 0 (0) | 3 (3)
Non-cardiac chest pain (Endocrine disorders) | 0 (0) | 3 (3)
Vision Blurred (Eye disorders) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 19 (19) | 11 (11)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 9 (9)
Vomiting (Gastrointestinal disorders) | 4 (4) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 5 (5)
Constipation (Gastrointestinal disorders) | 2 (2) | 5 (5)
Dry Mouth (Gastrointestinal disorders) | 5 (5) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 5 (5)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 3 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 3 (3)
Irritability (General disorders) | 3 (3) | 4 (4)
Disturbance in attention (General disorders) | 1 (1) | 3 (3)
Hypersensitivity (General disorders) | 1 (1) | 3 (3)
Upper Respiratory Tract Infection (Infections and infestations) | 8 (8) | 7 (7)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 25 (25) | 24 (24)
Sedation (Nervous system disorders) | 5 (5) | 8 (8)
Dizziness (Musculoskeletal and connective tissue disorders) | 7 (7) | 4 (4)
Migraine (Nervous system disorders) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 6 (6) | 11 (11)
Depression (Psychiatric disorders) | 2 (2) | 3 (3) — worse than baseline
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 8 (8)
Pruritis (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes